CLINICAL TRIAL: NCT01876173
Title: Development of and Feasibility Testing of Decision Support for Patients Who Are Candidates for an Implantable Defibrillator
Brief Title: Feasibility Testing of Decision Support for Patients Who Are Candidates for an Implantable Defibrillator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sandra Carroll, Assistant Professor, McMaster University
Allocation: Randomized | Model: Parallel | Purpose: Health Services Research
Other Study IDs: 12-214; 119449 Grant number (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2013-05-30; First posted 2013-06-12 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Disease; Sudden Cardiac Death
Keywords: Sudden cardiac death; implantable cardioverter defibrillator; decision aid
MeSH Terms: conditions — Cardiovascular Diseases; Death, Sudden, Cardiac | interventions — Primary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Decision Aid for an ICD (primary prevention, non-CRT) (Experimental): The intervention group will receive the PtDA, which provides a lay summary that outlines the facts, risks, benefits (including probabilities), specific to the option of an implantable defibrillator or the option of medical management to prepare them for consultation with the physician. Values are assessed to reveal which features of each option are important to patients.
  Interventions: Behavioral: Patient Decision Aid for an ICD (primary prevention, non-CRT)
- Usual care (No Intervention): The control group will not receive the patient decision aid prior to consultation with the physician.

INTERVENTIONS:
Behavioral: Patient Decision Aid for an ICD (primary prevention, non-CRT) — The intervention group will receive the PtDA, which provides a lay summary that outlines the facts, risks, benefits (including probabilities), specific to the option of an implantable defibrillator or the option of medical management to prepare them for consultation with the physician. Values are assessed to reveal which features of each option are important to patients.
  Other Names: PtDA
  Arms: Patient Decision Aid for an ICD (primary prevention, non-CRT)

SUMMARY:
Sudden cardiac death (SCD) due to a ventricular arrhythmia is a serious cause of cardiovascular death in Canada. The implantable cardioverter defibrillator (ICD) offers high-risk patients a treatment option to reduce the incidence of SCD by delivering an internal shock to restore a normal rhythm, if needed. Definitive evidence has established the effectiveness of the ICD for reducing mortality when used as prophylaxis for SCD (a primary prevention indication). Approximately 3,700 new candidates accrue annually. Practice guidelines define the criteria to determine patient ICD candidacy for primary prevention. However, in addition to SCD risk, ICD candidates may have chronic diseases such as diabetes, renal insufficiency, hypertension, and atrial fibrillation. Thus, balancing the benefits and risks of an ICD can become complex, particularly when competing mortality risks are present. Research has recognized human costs associated with device complications and shocks affecting psychological, health related quality of life (HRQL), and morbidity outcomes. The complexities surrounding the long-term benefits/risks, complications, replacements, and shocks, warrant decision support to prepare patients to make decisions. In Canada, there is no clear framework to support patients' decision-making in the context of ICD treatment options. Decision support, using a decision aid, could moderate treatment related uncertainty and prepare patients to make active, informed, quality decisions.

Objectives: 1) develop a decision aid for ICD candidates to support quality decision-making (informed, deliberate, values-based choices), 2) to evaluate the decision aid, and 3) to determine the feasibility of conducting a trial.

ELIGIBILITY:
Inclusion Criteria:

* Referred for consideration of an ICD(non-CRT)for a primary prevention indication
* English speaking
* able to provide informed consent

Exclusion Criteria:

* unable to understand the decision aid due to a language barrier or visual impairment
* referred for secondary prevention indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes(composite): i) decision aid development, and ii) decision aid evaluation. | Phase 1-2 (1- year)
  Development of the decision aid will be guided by the Ottawa Decision Support Framework (ODSF). Evaluation will include the Decision Aid Acceptability questionnaire comprised of 10 items including comprehensibility, balance of presentation of information, and overall suitability.

SECONDARY OUTCOMES:
Pilot RCT (feasibility) | Pre-Post consultation - participants will be followed until consultation is completed and at 3 months post consultation (average of 16 weeks)
  In this feasibility RCT, the feasibility regarding processes (referral and recruitment rates, consent), key to the success of a larger study will be assessed. This includes successful delivery of the decision aid in an efficient manner, the monitoring of resources (budget), and study management (trial coordination, human resources). We will assess the proportion of patients who complete the decision aid, quality questionnaires, and missing data.
Decision quality measures | Pre consultation (baseline visit)
  Decision quality, the extent to which patients' decisions are informed (knowledge) and values based (values, preferences, decisional conflict).
Decisional Conflict Scale (DCS) | Pre and post consultation- (intervention and usual care group, baseline visit + 1 week post consult)
  The Decisional Conflict Scale measures a person's perception of the difficulty in making a decision, the extent to which they feel uncertain about treatment options, are knowledgeable about the risks and benefits of options, clear about personal values, and supported in decision making. The scale has good test-retest reliability (Cronbach's alpha coefficients > 0.78) and predictive validity.
Sure Test | Pre-consultation - baseline visit
  The Sure Test is a 4 item decisional conflict screening tool designed for use in clinical practice. The Sure Test is embedded in the decision aid (intervention group).
The Center for Epidemiologic Studies Depression Scale (CES-D) | Pre consultation - baseline visit (intervention and usual care)
  The CES-D has 20 items that measure depressive symptoms. The CES-D has good reliability and validity across community and clinical settings. Associations between depressive symptoms and decision choice will be assessed.
Preparation for Decision Making scale | Post consultation - up to two weeks post baseline visit (intervention group)
  The Preparation for Decision Making Scale has 10 categorical items assessing the usefulness of the decision aid in preparing patients to communicate with a health professional.
The Medical Outcomes Trust Short Form (SF-36v2) | Pre consultation - baseline visit (intervention and usual care)
  The SF-36 is a reliable and valid generic health related quality of life scale (HRQL) comprised of 36 items. Associations between HRQL and decision choice will be undertaken.

OTHER OUTCOMES:
Vital status | 3 months post baseline visit
  Alive, deceased
Implant status | Phase 3, three months post baseline visit
  Device status - implantable defibrillator/no implantable defibrillator, deferred

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L Carroll, PhD, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Carroll SL, Stacey D, McGillion M, Healey JS, Foster G, Hutchings S, Arthur HM, Browne G, Thabane L. Evaluating the feasibility of conducting a trial using a patient decision aid in implantable cardioverter defibrillator candidates: a randomized controlled feasibility trial. Pilot Feasibility Stud. 2017 Nov 21;3:49. doi: 10.1186/s40814-017-0189-9. eCollection 2017. PMID 29201388
- [Derived] Carroll SL, McGillion M, Stacey D, Healey JS, Browne G, Arthur HM, Thabane L. Development and feasibility testing of decision support for patients who are candidates for a prophylactic implantable defibrillator: a study protocol for a pilot randomized controlled trial. Trials. 2013 Oct 22;14:346. doi: 10.1186/1745-6215-14-346. PMID 24148851
- See also: Related Info — http://decisionaid.ohri.ca/index.html